CLINICAL TRIAL: NCT02315573
Title: Lidocaine With Epinephrine vs. Bupivacaine With Epinephrine as Local Anesthetic Agents in Wide-awake Hand Surgery: an Outcome Study of Patients' Pain Perception.
Brief Title: Lidocaine With Epinephrine vs. Bupivacaine With Epinephrine as Local Anesthetic Agents in Wide-awake Hand Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Mary's Research Center, Canada (Other)
Responsible Party: Principal Investigator, Dr Mario Luc, Dr Mario Luc MD, MSc, FRCSC, St. Mary's Research Center, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMHC #14-30
Record Dates: First submitted 2014-12-03; First posted 2014-12-12 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Anesthetics, Local; Pain Perception; Pain Measurement; Analgesia; Lidocaine; Bupivacaine
MeSH Terms: conditions — Carpal Tunnel Syndrome; Agnosia | interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine with epinephrine (Experimental): Wrist block anesthesia with Lidocaine 1% with epinephrine; 10cc.
  Group 1 will receive the same treatment as group 2, except that the wide-awake carpal tunnel release surgery will be performed under Lidocaine anesthesia instead of Bupivacaine anesthesia.
  Interventions: Procedure: Wrist block anesthesia
- Bupivacaine with epinephrine (Experimental): Wrist block anesthesia with Bupivacaine 0.25% with epinephrine; 10cc.
  Group 2 will receive the same treatment as group 1, except that the wide-awake carpal tunnel release surgery will be performed under Bupivacaine anesthesia instead of Lidocaine anesthesia.
  Interventions: Procedure: Wrist block anesthesia

INTERVENTIONS:
Procedure: Wrist block anesthesia — The carpal tunnel release surgery will be performed under wrist block anesthesia. Group 1 will have the wrist block performed with Lidocaine and epinephrine, while Group 2 with Bupivacaine and epinephrine.
  Other Names: Lidocaine with epinephrine; Bupivacain with epinephrine

SUMMARY:
This study is focused on comparing patients' pain scores on a visual analogue scale (VAS) and the difference in analgesics use post-operatively (with the same prescription defining only the maximum frequency) between lidocaine with epinephrine & bupivacaine with epinephrine as local anesthetics in wide-awake hand surgery. The investigators' hypothesis states that a longer acting local anesthetic agent (bupivacaine) would be able to provide better postoperative pain relief demonstrated by lower pain scores on VAS and less analgesics use (as will be recorded on the patient's log). This will be mainly obvious in the first 24 hours postoperative period when the pain is usually at maximum levels and starts to decline thereafter. If the investigators' hypothesis is true, this may potentially change practices of many hand surgeons towards the routine use of longer acting local anesthetics particularly in wide-awake hand surgery, and perhaps could be extrapolated to other surgical specialties. Further, a reduction in postoperative analgesics use would be of paramount clinical importance, as it would reduce their potential side effects.

DETAILED DESCRIPTION:
The purpose of this study is to better understand the differences of two commonly used local anesthetics in carpal tunnel surgery. This study will explore the differences in terms of patient satisfaction during surgery (measured on VAS), pain after surgery (measured on VAS), and the need for pain medications after surgery (patients will annotate on a log given to them the time of the medication taken if needed for analgesia).

Wide awake hand surgery (freezing your limb while being fully awake) has recently been popularized as being faster and safer for patients compared to hand surgery under general anesthesia or with sedation. Advantages include fast recovery and no risks of general anesthesia.

In order to freeze the wrist to undergo carpal tunnel surgery, a local anesthetic is injected into the nerves of the wrist. Among the most commonly used anesthetic agents are Lidocaine (shorter duration of anesthesia) and Bupivacaine (longer duration of anesthesia). Until now, no enough evidence to support using one anesthetic agent over the other. Furthermore, no previous studies looked at the perception of pain from patient's perspectives when using different anesthetic agents.

There will be NO change in the standard medical care that patients will receive whether or not patients decide to participate in the study. Patients that join the study will receive the same anesthetic agents used in those procedures as patients who decide not to participate. The only difference will be collecting clinical data from participants and asking participants to complete two questionnaires regarding the surgical experience, and the perceived level of pain during the two days that follow surgery. As well, participants will be asked to keep a simple log of the pain medications that are consumed during the two days after the surgery. Patients' total participation time should take no more than 30 minutes.

Patients' decision to participate in this study will help doctors in the future to decide which of these two used anesthetic agents (Lidocaine or Bupivacaine) gives patients the best experience during surgery. As well, it will help reduce the pain that some patients experience after surgery, as well as reduce the need for pain medications after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* First time carpal tunnel surgery

Exclusion Criteria:

* Regular analgesic medication consumption
* More than one surgical procedure at the same time as carpal tunnel surgery
* Need for a surrogate decision maker
* Allergic or unable to take morphine, hydromorphone (Dilaudid), acetaminophen (Tylenol), lidoxaine (Xylocaine), bupivacaine (Marcane), or epinephrine
* End stage kidney disease
* End stage liver disease
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-10; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Pain scores on a visual analogue scale | 24 hours
  Patients' pain scores on a visual analogue scale over the first 24 hours after surgery.
Pattern and amount of analgesics consumed | 48 hours
  The time of consumption and the type of analgesic (acetaminophen 1g PO q6hr PRN or morphine 5mg PO q4hr PRN) consumed over the first 48 hours after surgery. This will be recorded in the medication log given to patients.

SECONDARY OUTCOMES:
Pain scores on a visual analogue scale | 24 hours
  Patients' pain scores on a visual analogue scale perceived between the first 24 hours and 48 hours after surgery.
Patient satisfaction scores on a visual analogue scale | Immediate
  Patient self rated satisfaction on a visual analogue scale with wide-awake carpal tunnel release surgery. Will be measured immediately after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Luc, MD, FRCSC, Principal Investigator — McGill University
Locations (1):
- St. Mary's Hospital Center, Montreal, Quebec, Canada

REFERENCES:
- [Background] Wildin C, Dias JJ, Heras-Palou C, Bradley MJ, Burke FD. Trends in elective hand surgery referrals from primary care. Ann R Coll Surg Engl. 2006 Oct;88(6):543-6. doi: 10.1308/003588406X117070. PMID 17059713
- [Background] Angermann P, Lohmann M. Injuries to the hand and wrist. A study of 50,272 injuries. J Hand Surg Br. 1993 Oct;18(5):642-4. doi: 10.1016/0266-7681(93)90024-a. PMID 8294834
- [Background] Larsen CF, Mulder S, Johansen AM, Stam C. The epidemiology of hand injuries in The Netherlands and Denmark. Eur J Epidemiol. 2004;19(4):323-7. doi: 10.1023/b:ejep.0000024662.32024.e3. PMID 15180102
- [Background] Neill RS. Postoperative analgesia following brachial plexus block. Br J Anaesth. 1978 Apr;50(4):379-82. doi: 10.1093/bja/50.4.379. PMID 656255
- [Background] Ganzberg S, Kramer KJ. The use of local anesthetic agents in medicine. Dent Clin North Am. 2010 Oct;54(4):601-10. doi: 10.1016/j.cden.2010.06.001. PMID 20831924
- [Background] Alhelail M, Al-Salamah M, Al-Mulhim M, Al-Hamid S. Comparison of bupivacaine and lidocaine with epinephrine for digital nerve blocks. Emerg Med J. 2009 May;26(5):347-50. doi: 10.1136/emj.2008.062497. PMID 19386869
- [Background] Conolly WB, Berry FR. The place of peripheral nerve blocks in reconstructive hand surgery. Hand. 1977 Jun;9(2):157-9. doi: 10.1016/s0072-968x(77)80011-9. PMID 914091
- [Background] Lalonde DH. Reconstruction of the hand with wide awake surgery. Clin Plast Surg. 2011 Oct;38(4):761-9. doi: 10.1016/j.cps.2011.07.005. PMID 22032599
- [Background] Pratap JN, Shankar RK, Goroszeniuk T. Co-injection of clonidine prolongs the anesthetic effect of lidocaine skin infiltration by a peripheral action. Anesth Analg. 2007 Apr;104(4):982-3. doi: 10.1213/01.ane.0000257949.46444.a8. PMID 17377118
- [Background] Reinhart DJ, Stagg KS, Walker KG, Wang WP, Parker CM, Jackson HH, Walker EB. Postoperative analgesia after peripheral nerve block for podiatric surgery: clinical efficacy and chemical stability of lidocaine alone versus lidocaine plus ketorolac. Reg Anesth Pain Med. 2000 Sep-Oct;25(5):506-13. doi: 10.1053/rapm.2000.7624. PMID 11009237
- [Background] Thomson CJ, Lalonde DH. Randomized double-blind comparison of duration of anesthesia among three commonly used agents in digital nerve block. Plast Reconstr Surg. 2006 Aug;118(2):429-32. doi: 10.1097/01.prs.0000227632.43606.12. PMID 16874214
- [Background] Reichl M, Quinton D. Comparison of 1% lignocaine with 0.5% bupivacaine in digital ring blocks. J Hand Surg Br. 1987 Oct;12(3):375-6. doi: 10.1016/0266-7681_87_90192-6. PMID 3325593
- [Background] Gorzack A. Towards evidence based emergency medicine: best BETs from the Manchester Royal Infirmary. Lignocaine or bupivacaine for digital ring block. J Accid Emerg Med. 1998 Sep;15(5):353. doi: 10.1136/emj.15.5.353. No abstract available. PMID 10454811
- [Background] Valvano MN, Leffler S. Comparison of bupivacaine and lidocaine/bupivacaine for local anesthesia/digital nerve block. Ann Emerg Med. 1996 Apr;27(4):490-2. doi: 10.1016/s0196-0644(96)70239-1. PMID 8604868
- [Background] Nystrom A, Lindstrom G, Reiz S, Hanel DP. Bupivacaine: a safe local anesthetic for wrist blocks. J Hand Surg Am. 1989 May;14(3):495-8. doi: 10.1016/s0363-5023(89)80010-3. PMID 2544640
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Background] Shrout PE, Fleiss JL. Intraclass correlations: uses in assessing rater reliability. Psychol Bull. 1979 Mar;86(2):420-8. doi: 10.1037//0033-2909.86.2.420. PMID 18839484